CLINICAL TRIAL: NCT05173363
Title: Influence of Square-stepping Exercise on Brain Activation, Cognitive Function and Physical Performance in Frail Elders With MCI
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: YM110152F
Record Dates: First submitted 2021-12-05; First posted 2021-12-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2022-09

CONDITIONS: Frailty; Mild Cognitive Impairment
Keywords: Square-stepping exercise; Frailty; Mild Cognitive Impairment
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults with frailty and mild cognitive impairment

SUMMARY:
This study is to elucidate the possible mechanisms of SSE by examining brain activation differences between SSE patterns and usual walking, as well as the relationship between brain activity and SSE performance, between cognitive function and SSE performance, and between physical performance and SSE performance in frail elders with MCI.

DETAILED DESCRIPTION:
Background:

Both frailty and MCI exert negative impact on motor and cognitive function, which increase the risks of fall and adverse health condition. SSE has been proved to be an effective intervention for motor and cognitive function in older adults. However, the underlying mechanisms of SSE still remain undetermined for its possible effects. This study aims to elucidate the possible mechanisms of SSE in frail elders with MCI.

Methods:

This is a cross-sectional study. The inclusion criteria are: (1) age between 65 and 90 years old, (2) the presence of at least 1 characteristic of the Fried frailty criteria, (3) with mini-mental state examination (MMSE) score≧24 and Montreal Cognitive Assessment (MoCA) score <26 (MCI criteria), and (4) ability to walk independently for 1 min without assistive devices. The exclusion criteria are: (1) central nervous system disorders (such as stroke, Parkinson's disease, spinal cord injury), and (2) any unstable physical condition, psychiatric disorder, and other neurological disorder or diagnosed with learning disability which may affect participating this study. Brain activity during SSE and usual walking, SSE performance, physical performance, and cognitive function are measured. The purpose of this study is to elucidate the possible mechanisms of SSE by examining brain activation differences between SSE patterns and usual walking, as well as the relationship between brain activity and SSE performance, between cognitive function and SSE performance, and between physical performance and SSE performance in frail elders with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 90 years old
* Presence of at least 1 characteristic of the Fried frailty criteria
* Mini-mental state examination score equal to or more than 24
* Montreal Cognitive Assessment score less than 26
* Ability to walk independently for 1 min without assistive devices

Exclusion Criteria:

* Central nervous system disorders (such as stroke, Parkinson's disease, spinal cord injury)
* Any unstable physical condition, psychiatric disorder, and other neurological disorder or diagnosed with learning disability which may affect participating this study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults with frailty and mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Brain activity | 20 minutes
  The brain activity will be measured under 3 tasks: usual walking, SSE-pattern1 (SSE1), and SSE-pattern 2 (SSE2)
SSE performance | 15 minutes
  The number of the correct steps that participants complete in 1 min during SSEs will be recorded
Montreal Cognitive Assessment | 15 minutes
  Global cognitive function
Trail making test | 5 minutes
  Executive function
Stroop color and word test | 5 minutes
  Executive function
Digit span test | 8 minutes
  Executive function
Timed up and go test | 5 minutes
  Dynamic balance and functional mobility
Berg balance scale | 15 minutes
  Balance and fall risk
Five times sit to stand test | 3 minutes
  Lower extremity strength

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No